CLINICAL TRIAL: NCT05046808
Title: A Single-center, Randomized, Open-label Pharmacokinetic Study of Famitinib Malate Capsules in Healthy Subjects
Brief Title: Pharmacokinetics Study of Famitinib Malate Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FMTN-I-110
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Famitinib Malate Capsules 10mg (Experimental)
  Interventions: Drug: Famitinib Malate Capsules
- Famitinib Malate Capsules 15mg (Experimental)
  Interventions: Drug: Famitinib Malate Capsules
- Famitinib Malate Capsules 20mg (Experimental)
  Interventions: Drug: Famitinib Malate Capsules
- Famitinib Malate Capsules 10mg*2 (Experimental)
  Interventions: Drug: Famitinib Malate Capsules
- Famitinib Malate Capsules 25mg (Experimental)
  Interventions: Drug: Famitinib Malate Capsules

INTERVENTIONS:
Drug: Famitinib Malate Capsules — Famitinib Malate Capsules 10mg single dose
  Arms: Famitinib Malate Capsules 10mg
Drug: Famitinib Malate Capsules — Famitinib Malate Capsules 15mg single dose
  Arms: Famitinib Malate Capsules 15mg
Drug: Famitinib Malate Capsules — Famitinib Malate Capsules 20mg single dose
  Arms: Famitinib Malate Capsules 20mg
Drug: Famitinib Malate Capsules — Famitinib Malate Capsules 10mg*2 single dose
  Arms: Famitinib Malate Capsules 10mg*2
Drug: Famitinib Malate Capsules — Famitinib Malate Capsules 25mg single dose
  Arms: Famitinib Malate Capsules 25mg

SUMMARY:
This is a single-center, randomized, open-label study to compare the pharmacokinetic profiles of Famitinib and its metabolite SHR116637 at different doses/specifications.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: healthy male and female subjects.
2. Age: 18 years old and above (including 18 years old).
3. Weight: male subjects should not be less than 50.0kg, female subjects should not be less than 45.0kg, body mass index [BMI=weight (kg)/height2 (m2)] is 19.0 to 26.0kg/m2 (including boundary values).
4. Subjects with fertility and their partners have no fertility plan and voluntarily take medically approved high-efficiency contraception methods (see appendix 1 for details), and no plan to donate eggs or sperm within 28 weeks after signing the informed consent. Women with childbearing potential must have a negative serum pregnancy test within 24 hours before taking the study drug for the first time.
5. Subjects must give informed consent to this study before the experiment, and voluntarily sign a written informed consent form.
6. The subject can communicate well with the researcher and can complete the research in accordance with the research regulations.

Exclusion Criteria:

1. Those who are allergic to the active ingredients of the preparation and related compounds and any excipients or are allergic to two or more drugs (or food).
2. Those who cannot follow a unified diet (such as intolerance to standard meals, etc.).
3. Those who cannot tolerate venepuncture, and those who have a history of fainting needles and bleeding.
4. There is a history of cardiovascular (such as hypertension), liver, kidney (such as chronic kidney disease), endocrine, blood system, respiratory system, malignant tumour, mental abnormality, severe infection, etc. or the existing above diseases that the researcher judges to be clinically significant.
5. Chronic or active gastrointestinal diseases such as esophagitis, gastritis, gastric ulcer, enteritis, gastrointestinal bleeding, gastroesophageal reflux disease, gastrointestinal obstruction, oesophageal varices, or gastrointestinal surgery (part of the digestive tract resection, cholecystectomy), etc., and the investigator believes that there is still clinical significance.
6. During the screening period, there are serious gastrointestinal symptoms (such as nausea, vomiting, stomach pain, abdominal pain, diarrheal, abdominal discomfort, abdominal distension, etc.), and the investigator believes that it is currently clinically meaningful.
7. Patients with upper respiratory tract infection during the screening period, and the investigator believes that it is currently clinically significant.
8. Those who have undergone major surgery within 6 months before screening, or who plan to undergo surgery during the study period, and those who have undergone surgery that will affect drug absorption, distribution, metabolism, and excretion (except for appendicitis surgery).
9. During the screening period, physical examination, vital signs, 12-lead electrocardiogram, chest radiograph, abdominal ultrasound, blood routine, blood biochemistry, urine routine, blood coagulation and thyroid function (FT3, FT4, TSH) abnormalities, the investigator judged that the abnormalities have clinical significance.
10. Abnormal test results of hepatitis B surface antigen, hepatitis C virus antibody, Treponema pallidum antibody or human immunodeficiency virus antibody have clinical significance.
11. Those who drank excessive amounts of tea, coffee, or caffeinated beverages (more than 8 cups a day, 1 cup = 200 mL) within 3 months before screening; or consumed any food or beverages containing caffeine within 48 hours before the first administration of the study drug (Such as coffee, strong tea, chocolate, etc.).
12. Those who have consumed any beverages or foods that are rich in xanthine or grapefruit ingredients or other beverages or foods that affect the absorption, distribution, metabolism, and excretion of the drug within 48 hours before the first administration of the study drug.
13. Any drug that interacts with this drug has been used within 4 weeks before screening (see appendix 3).
14. Those who have used long-acting estrogen or progestin injections or implants within 6 months before the test; those who have used short-acting contraceptives within 30 days before the test.
15. Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health care products in the 14 days before the first administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for Famitinib after Single dose | from Day 1 to Day 9 after the first dose
Area under the plasma concentration versus time curve (AUC0-t) for Famitinib after Single dose | from Day 1 to Day 9 after the first dose
Area under the plasma concentration versus time curve (AUC0-∞) for Famitinib after Single dose | from Day 1 to Day 9 after the first dose
Time to maximum observed plasma concentration (Tmax) for Famitinib after Single dose | from Day 1 to Day 9 after the first dose
Elimination half-life (T1/2) for Famitinib after Single dose | from Day 1 to Day 9 after the first dose
Apparent oral clearance (CL/F) for Famitinib after Single dose | from Day 1 to Day 9 after the first dose
Apparent Volume of Distribution (Vz/F) Famitinib after Single dose | from Day1 to Day9 after the first dose
Maximum observed plasma concentration (Cmax) for SHR116637 after Single dose | from Day 1 to Day 9 after the first dose
Area under the plasma concentration versus time curve (AUC0-t) for SHR116637 after Single dose | from Day 1 to Day 9 after the first dose
Area under the plasma concentration versus time curve (AUC0-∞) for SHR116637 after Single dose | from Day 1 to Day 9 after the first dose
Time to maximum observed plasma concentration (Tmax) for SHR116637 after Single dose | from Day 1 to Day 9 after the first dose
Time to elimination half-life (T1/2) for SHR116637 after Single dose | from Day 1 to Day 9 after the first dose
Apparent oral clearance (CL/F) for SHR116637 after Single dose | from Day 1 to Day 9 after the first dose
Apparent Volume of Distribution (Vz/F) SHR116637 after Single dose | from Day 1 to Day 9 after the first dose

SECONDARY OUTCOMES:
Number of subjects with adverse events and severity of adverse events | from Day 1 to Day 16 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided